CLINICAL TRIAL: NCT04408170
Title: Facilitating AcceLerated Clinical Validation Of Novel Diagnostics for COVID-19 (FALCON-C19)
Acronym: FALCON-C19
Status: Completed | Type: Observational
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: B00944
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Coronavirus Infection; COVID-19
Keywords: In vitro diagnostics; Point-of-care testing
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Throat and nose swabs and/or saliva samples may be taken at multiple time points and stored for future testing.
  Whole blood samples may be taken at multiple time points during the study. Samples will be processed and the serum stored.
  Finger stick samples may also be taken and stored for future testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Work Stream A: Patients that are recruited in hospital with either query COVID-19 or who have tested positive for COVID-19.
  Interventions: Diagnostic Test: Point-of-care test for SARS-CoV-2
- Work Stream B: Known COVID-positive and/or COVID-negative community testing
  Interventions: Diagnostic Test: Point-of-care test for SARS-CoV-2
- Work Stream C: Undifferentiated community testing
  Interventions: Diagnostic Test: Point-of-care test for SARS-CoV-2

INTERVENTIONS:
Diagnostic Test: Point-of-care test for SARS-CoV-2 — Throat and nose swabs and/or saliva samples and/or whole blood and/or finger stick samples may be taken to be tested on Point-of-care tests for SARS-CoV-2

SUMMARY:
The United Kingdom and wider world is in the midst of the 2019 novel coronavirus (SARS-CoV-2) pandemic. Accurate diagnosis of infection, identification of immunity and monitoring the clinical progression of infection are of paramount importance to our response. Widespread population testing has proven difficult in western countries and has been limited by test availability, human resources and long turnaround times (up to 72 hours). This has limited our ability to control the spread of infection and to develop effective clinical pathways to enable early social isolation of infected patients and early treatment for those most at risk. The life sciences industry has responded to the pandemic by developing multiple new in vitro diagnostic tests (IVDs). To leverage the potential clinical benefit of those tests we require efficient but robust clinical evaluation. Therefore, to optimise resource utilisation in this global pandemic, we will conduct a platform adaptive diagnostic study on a national level, utilising a national network of expertise in the evaluation of diagnostic technology. This study will enable the evaluation of multiple assays in three priority areas:

1. Evaluation of the diagnostic accuracy of IVDs for active infection with SARS-CoV-2
2. Evaluation of assays monitoring the immune response to SARS-CoV-2 infection
3. Evaluation of the prognostic value of commercially available tests for predicting prognosis in patients with suspected or confirmed SARS-CoV-2 infection. (This arm will not be active immediately but may be activated after initiation).

ELIGIBILITY:
Work Stream A (in-hospital; Group 1 and Group 2):

Group 1 Inclusion Criteria:

We will include participants (patients or staff):

1. That are 18 years or older
2. That will require testing for COVID-19 in the opinion of the treating clinician
3. That may have presented with acute symptoms of COVID-19 (e.g. fever, cough, dyspnoea, anosmia) or chest x-ray changes or they may be asymptomatic but require testing for other reasons

Group 2 Inclusion Criteria:

We will include participants:

1. That are 18 years or older
2. That have been admitted for another reason other than suspected SARS-CoV-2 infection, but when routinely swabbed they have been identified as positive for SARS-CoV-2 PCR

Work Stream B (Group 3):

We will include participants:

1. That are 18 years or older

   EITHER:
2. They have been identified as positive for SARS-CoV-2 PCR through testing at national laboratory infrastructure OR
3. They have been identified as negative for SARS-CoV-2 PCR through testing at national laboratory infrastructure

Work Stream C (Group 4):

We will include participants:

1. That are 18 years or older
2. Who are undergoing testing for COVID-19, whether they are symptomatic or symptomatic for COVID-19

Exclusion Criteria for all Work Streams:

1. Patients where it is impossible/unsafe to obtain the required research samples
2. Prisoners
3. Patients where sampling is not feasible

Ages: 18 Years to 100 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Work Stream A: Patients who present or are referred to secondary/tertiary care settings due to possible SARS-CoV-2 infection
  Work Stream B: Known COVID-positive and/or COVID-negative community testing
  Work Stream C: Undifferentiated community testing
Sampling Method: Non-Probability Sample
Enrollment: 8380 (Actual)
Dates: Start 2020-05-19 (Actual); Primary Completion 2021-01-26 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
If the participant has an active SARS-CoV-2 infection during admission | Baseline
  This will be determined using the point-of-care test and the laboratory test results
The participant has had a past SARS-CoV-2 infection | Day 90
  This will be determined using the point-of-cacre test for SARS-CoV-2 antibodies and the laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Richard Body, Study Director — Manchester University NHS Foundation Trust
Locations (15):
- United Kingdom (15):
  - Sandwell General Hospital Birmingham NHS Trust, Birmingham
  - University Hospitals of Derby and Burton NHS FT, Derby
  - Frimley Health NHS FT, Frimley
  - Airedale NHS FT, Keighley
  - Leeds Teaching Hospital NHS FT, Leeds
  - St George's University Hospitals NHS FT, London
  - Manchester University NHS FT, Manchester
  - Newcastle upon Tyne Hospitals NHS FT, Newcastle upon Tyne
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Oxford University Hospitals NHS FT, Oxford
  - Royal Berkshire Hospital NHS FT, Reading
  - Barking, Havering & Redbridge Hospitals NHS FT, Romford
  - Salford Royal NHS FT, Salford
  - University Hospital Southampton NHS FT, Southampton
  - University Hospitals of North Midlands NHS Trust, Stoke-on-Trent

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Byrne RL, Aljayyoussi G, Kontogianni K, Clerkin K, McIntyre M, Wardale J, Williams CT, Body R, Adams ER, de Vos M, Escadafal C, Cubas Atienzar AI. Head-to-head comparison of anterior nares and nasopharyngeal swabs for SARS-CoV-2 antigen detection in a community drive-through test centre in the UK. BMJ Open Respir Res. 2025 Mar 22;12(1):e001747. doi: 10.1136/bmjresp-2023-001747. PMID 40122534